CLINICAL TRIAL: NCT06595316
Title: A Randomized Controlled Feasibility Trial of a Vigorous Intensity Aerobic Exercise and Resistance Training Intervention for Mitigating Chemotherapy Cardiotoxicity in Breast Cancer Patients
Brief Title: Exercise for Ameliorating Chemotherapy Cardiotoxicity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RS216 - 338687
Record Dates: First submitted 2024-04-25; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiotoxicity
Keywords: exercise; cardiotoxicity; exercise oncology; breast cancer
MeSH Terms: conditions — Cardiotoxicity; Motor Activity; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants recruited will be cancer patients who attend to the Queen's Centre for Oncology and Haematology at Castle Hill Hospital, whose confirmed diagnosis is ER+ HER2- breast cancer, and whose chemotherapy regimen is 3 cycles of epirubicin and cyclophosphamide (EC) followed by 3 cycles docetaxel over a period of 18 weeks. They will be identified, screened and selected according to the study's inclusion and exclusion criteria, and then approached by their Consultant Clinical Oncologist in charge and/or the researcher. Patients will be offered the opportunity to be part of the study. Individuals will only participate if they have provided informed consent.
  Participants will be randomly allocated in a 1:1 ratio, either to intervention group, or the control group (usual care) by an unrestricted simple random sampling technique, until the maximum number of participants has been reached, which is a total of 15 individuals per group over a period of maximum 15 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise intervention group (Experimental): For this group (N=15) the intervention will consist of two supervised sessions per week, which include aerobic and resistance exercise, carried out as previuosly described.
  Interventions: Other: Exercise intervention group
- Control group (usual care) (No Intervention): For the Control group or usual care (N=15), there will be no exercise sessions. Although, the same assessments as the intervention group will be carried out, at the same time-points.

INTERVENTIONS:
Other: Exercise intervention group — Exercise will consist of two supervised sessions per week. Starting with vital signs monitoring (blood pressure, temperature, blood oxygen levels, heart rate).
  The aerobic component consists of a 5-minute warm-up, followed by 3 bouts of 4-minute cycling at an intensity of 60-65% HRR, with 2-minute active recovery periods in between and a 5-minute cool down. The goal is to increase up to an intensity of around 80%-85% HRR by weeks 16 to 18. Intensity will be monitored with The Borg Rating Scale of Perceived Exertion (RPE). The resistance component will consist of upper body and lower body exercises (door frame rows, wall push-ups, glute bridges, triceps lifts and squat to calf rise) starting on week one with a set of 12 repetitions of each exercise, with 2-minute recovery in between exercises aiming to increase the number of sets and reducing the number of repetitions.
  Arms: Exercise intervention group

SUMMARY:
Chemotherapy is a common treatment for breast cancer but can damage the heart and blood vessels. Exercise, such as cycling, may stop chemotherapy from damaging the heart and blood vessels. Before the effects of exercise on the heart and blood vessels can be fully determined in a large trial, a small trial must first be carried out to assess if exercise can be included safely and practically during chemotherapy treatment.

This study is designed so that a group of breast cancer patients will exercise during their chemotherapy treatment, whilst another group does not exercise. Participants will be breast cancer patients from the Queen's Centre for Oncology and Haematology at Castle Hill Hospital. Suitable patients will be identified and approached by their Consultant Clinical Oncologist. If patients decide to take part, they will be randomly placed into groups ('exercise' or 'usual care') before starting chemotherapy. The exercise group will exercise for 50-60 minutes 2days/week in the Cardiac Rehabilitation Gym at Castle Hill Hospital during their chemotherapy treatment. Exercise will be supervised, consisting of repeated 5-minute bouts of high intensity cycling plus strength training. The usual care group will be given their normal chemotherapy only (no exercise). Both groups will take part in tests before they begin chemotherapy treatment. Tests assess heart and blood vessel health, fitness, strength, fatigue, and quality of life. The same tests will happen again during the intervention, after the intervention and 3-months later. Participants will also have to complete questionnaires to give their opinion of the study. The main point of the study is to determine if the exercise and tests are received well by patients, if recruitment is good, and if patients comply/adhere. This will inform a larger study which will assess if exercise maintains heart and vessel health during chemotherapy treatment.

DETAILED DESCRIPTION:
Exercise has been shown to have benefits within cardio-oncology settings and evidence supports the use of exercise as a cardioprotective method in breast cancer. Several studies demonstrate evidence for positive effects of aerobic and resistance exercise to improve or alleviate the usual effects of chemotherapy on the heart and blood vessels in breast cancer. Despite the existing evidence that shows promising outcomes regarding exercise interventions for breast cancer patients undergoing chemotherapy who are at risk of developing cardiotoxicity due to treatment there is still insufficient evidence for exercise to be prescribed to this population as an adjuvant instrument to reduce cardiotoxicity.

Through this study we aim to build on the evidence base with the purpose of encouraging practice towards this approach. However, before a large definitive randomized controlled trial (RCT) can be conducted, the first step is to assess the feasibility of a high intensity exercise intervention during chemotherapy for breast cancer. This will inform the design of a large RCT which will determine the cardio-protective effects of the exercise intervention.

As this is a feasibility study the main outcome is to find out the practicalities of delivering the proposed exercise intervention in a healthcare setting by collecting information regarding eligibility, recruitment rates, retention, adherence, fidelity, and adverse events.

Secondary outcome measures will provide information about cardiac function, cardiovascular toxicity and inflammation, electrical activity of the heart, vascular function, functional capacity, muscle strength, fatigue, quality of life, and finally experiences and perceptions of patients after participating in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 to 75 years old.
* Confirmed early stage (I-III) ER+ HER2 - breast cancer diagnosis
* Undergoing adjuvant and neoadjuvant chemotherapy, consisting of epirubicin and cyclophosphamide (EC) followed by Docetaxel.
* No contraindications to engage in physical activity.
* Capable of giving informed consent.
* Patients able to understand and communicate in English language

Exclusion Criteria:

* Participants with cognitive disorders
* Cancer metastases
* Uncontrolled or serious illnesses that might hamper patients' capacity of exercising

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Feasibility Log of Eligibility of Participants. | Eligibility will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Eligibility of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information regarding the number of patients able to take part of the study after shared characteristics as a population have been assessed.
Quantitative Feasibility Log of Recruitment of Participants | Recruitment will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Recruitment of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information considering the number of randomized patients over the total number of months of recruitment time.
Quantitative Feasibility Log of Retention of Participants | Retention will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Retention of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information where Retention will be assessed by the formula based on the number of participants at the end of the set time period divided by the number of patients participating at the start of the set time period and multiplied by 100.
Quantitative Feasibility Log of Attendance of Participants | Retention will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Attendance of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information regarding the number of sessions attended per each patient, throughout the program.
Quantitative and Qualitative Feasibility Log of Adverse Events of Participants | Adverse Events will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Adverse Events of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative and qualitative information regarding details of reactions to the exercise intervention like any cardiorespiratory complications, musculoskeletal injury or pain or discomfort.
Quantitative Feasibility Checklist of Fidelity | Fidelity will be recorded will be recorded during the weeks of exercise intervention, (18 weeks).
  To assess the feasibility of Intervention Fidelity of delivering the protocol to breast cancer patients undergoing chemotherapy. This will be measured by Checklist of Fidelity e.g., if exercise sessions start on time, if patients complete the exercise session, if exercise sessions finish on time. Every item is rated on binary metric where "0" equates No and "1" equates yes.
Quantitative Feasibility Log of Adherence of Participants | Adherence will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Adherence of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information regarding the percentage of classes attended out of the sessions planned.
Quantitative Feasibility Log of Compliance (duration) of Participants | Compliance will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Compliance of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by the total number of minutes per exercise session achieved over all weeks of the exercise programme (duration); this quantitative information will be recorded at the Researchers Log.
Quantitative Feasibility Log of Compliance (intensity) of Participants | Compliance will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Compliance of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by the intensity achieved by the patients during the intervention (%HRR); this quantitative information will be recorded at the Researchers Log.
Quantitative Feasibility Log of Completion (retention) of Participants | Completion (retention) will be recorded through study completion, an average of 15 months.
  To assess the feasibility of Completion (retention) of delivering the prescribed exercise protocol to breast cancer patients undergoing chemotherapy. This will be measured by a Researchers Log which will include quantitative information regarding the percentage of patients continuously attending and assessed at follow-up.
Qualitative Feasibility Log of Perception and experience of Participants | Perception and experience of Participants will be recorded within one week after the last exercise session of each patient has taken place.
  To assess the feasibility of the exercise protocol to breast cancer patients undergoing chemotherapy, Perception and experience of participants, as well as details of the impact this intervention had on their lives.will be recorded through an open-ended questions questionnaire. Information obtained will be recorded on the Researches Log.

SECONDARY OUTCOMES:
Echocardiographic scans - Left Ventricular Ejection Fraction (LVEF) | These assessments will be performed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  The Percentage of Left Ventricular Ejection Fraction (LVEF) will be measured as an outcome measure for cardiac function.
Echocardiographic scans - Peak systolic global longitudinal strain (GLS) | These assessments will be performed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  The percentage of Peak systolic global longitudinal strain (GLS) will be measured as an outcome measure for cardiac function.
Blood-borne biomarkers - Concentration of B-type natriuretic peptide (NT-ProBNP), Troponin I & T in blood samples. | These assessments will be performed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  B-type natriuretic peptide (NT-ProBNP), Troponin I & T will be measured,these are blood markers of cardiovascular toxicity and inflammation.
12-lead Electrocardiogram (ECG) | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  This assessment will help measure the electrical activity of the heart. Parameters considered will be: measurements (Heart Rate, PR Interval, QRS Duration, QT Interval, Frontal Plane QRS Axis), Rhythm (if normal or abnormal, P waves), Conduction (Normal Sino-atrial, Atrio-ventricular, and Intraventricular conduction, PR interval and QRS duration), Waveform Description, P Wave (P duration, P amplitude, Frontal plane P wave axis), QRS Complex (duration, amplitude, Frontal plane leads, Precordial leads), and ST Segment and T wave
Brachial artery flow-mediated dilation (FMD) | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  This test will be used to assess endothelium-dependent vasodilation, providing information about vascular function.
Aortic Pulse Wave Velocity (PWV) | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  This test will be used to assess vascular function since it enables the direct assessment of aortic stiffness.
The six Minute Walking Test (6MWT) | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  This assessment will be an outcome measure for patients' functional capacity.
Hand-grip Dynamometry | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  To assess muscle strength
30 seconds Sit-to-stand Tests | This will be assessed at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30).
  To assess muscle strength
The Functional Assessment of Chronic Disease Therapy | It will be completed by the participants at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30)
  To measure self-reported fatigue and how it affects daily life in patients. It consists of a 13-item questionnaire, every item is rated on a scale of 0 to 4. The higher the result, the more fatigue the patient presents.
The Functional Assessment of Cancer Therapy - Breast | It will be completed by the participants at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30)
  To examine the impact of health status on the quality of life. It is a 37-item instrument which measures five domains of Health Related Quality of Life (HRQOL) in breast cancer patients: Physical, social, emotional, functional well-being as well as a breast-cancer subscale (BCS); every item is rated on a scale of 0 to 4. The higher the result, the lower the HRQOL.
The 7-day Physical Activity Recall Scale | It will be completed by the participants at baseline (week 0), within one week after the last exercise session of each patient has taken place (week 19), and 3 months after the last exercise session of each patient has taken place (week 30)
  Is semi-structured questionnaire to estimate the individual's time spent in physical activity, strength, and flexibility activities for the last 7 days, allowing calculation of total energy expenditure and time spent in moderate, hard and very hard physical activity in units of energy which are metabolic equivalents (METs). The higher the mets, the higher the greater the amount of physical activity performed.

IPD SHARING:
Plan to Share IPD: No